CLINICAL TRIAL: NCT02126683
Title: The Effect of Plaquenil on Serum Inflammatory Markers and Goiter in Euthyroid Young Women With Hashimoto's Thyroiditis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201312121MINA
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Hashimoto's Thyroiditis
Keywords: Hashimoto's thyroiditis; Plaquenil
MeSH Terms: conditions — Hashimoto Disease | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plaquenil first (Experimental): Start Plaquenil 200mg BID orally since enrollment Duration: 6 months
  Interventions: Drug: Hydroxychloroquine
- Plaquenil later (Experimental): Start Plaquenil 200mg BID orally since the 25th week after enrollment Duration: 6 months
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine
  Other Names: Plaquenil

SUMMARY:
Hashimoto's thyroiditis (HT) is a common form of autoimmune thyroid disease, which affects up to 2% of general population. The annual incidence of HT worldwide is estimated to be 0.8 - 3.5 cases per 1000 persons. The thyroid gland attacked by a variety of cell- and antibody-mediated immune processes. Various auto-antibodies may be present against TPO and Tg, and ADCC is a substantial factor behind the apoptotic fall-out of HT. Activation of cytotoxic T-lymphocytes in response to cell-mediated immune response affected by helper T-cells is central to thyrocyte destruction. Recent studies showed higher pro-inflammatory cytokines in serum of patients with HT, and suggested HT is associated with regulatory T-cells dysfunction, imbalance of ratio of Th1 cell and Th2 cell, overexpression of Th17 cells.

Several studies suggested that pregnant women with HT, even at euthyroid state had higher risk of spontaneous miscarriage, more frequent post-partum depression and higher depressive, anger, and total mood disturbance risk compared to those without HT. Presence of thyroid auto-antibodies is also associated with negative pregnant outcomes including gestational hypertension, late abortion, fetal death, premature delivery and neonatal respiratory distress. Neonates from mothers with ATD have higher rate of transient hypothyroidism. Children of mothers with ATD had higher risk of positive serum thyroid auto-antibodies and development of goiter and thyroid dysfunction. However, there is no suggested treatment for subjects with HT who have normal thyroid function. Low-iodine diet and regularly follow-up were suggested.

Plaquenil (hydroxychloroquine) is an anti-malarial agent, and has been used to treat several autoimmune diseases, including lupus erythematosus and rheumatoid arthritis for more than a century. It reduced lymphocytes, production of auto-antibodies, cytokines, and immune mediators, NK cell activity, and inhibits antigens presenting to CD4 T-cells of B cells, dendritic cells and monocytes.

This study focuses on the effect of Plaquenil on thyroid auto-antibodies, inflammatory markers, cytokines, and goiter size in euthyroid women with HT.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed (within 1 year) Hashimoto's thyroiditis by positive serum anti-TPO antibody or anti-thyroglobulin antibody
* Euthyroid state by serum free T4 and TSH level within normal limit

Exclusion criteria:

* Pregnant, planning pregnant within 1 year, or lactating women
* Renal insufficiency, abnormal liver function test
* Hematologic diseases: anemia, agranulocytosis, thrombocytopenia
* G6PD deficiency, porphyria cutaneous tarda
* Allergy to 4-aminoquinoline compounds
* Known retinopathy or visual field defect disorders
* Already receive immunosuppression therapy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change of thyroid auto-antibodies | Baseline, up to 18 months
  Change of serum thyroid autoantibodies including anti-TPO antibody and anti-thyroglobulin antibody at baseline, and every 3 months after treatment intervention up to 18 months

SECONDARY OUTCOMES:
Change of inflammatory markers | Baseline, up to 18 months
  Change of serum inflammatory markers, including hsCRP and ESR at baseline, and every 3 months after treatment intervention up to 18 months
Change of proinflammatory markers | Baseline, up to 18 months
  Change of serum proinflammatory markers and cytokine level at baseline, and every 3 months after treatment intervention up to 18 months
Change of goiter size | Baseline, up to 18 months
  Change of thyroid volume measured by ultrasound at baseline, and every 3 months after treatment intervention up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Shang Huang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan